CLINICAL TRIAL: NCT04723121
Title: Can We Predict of the Response of High Risk Non Muscle Invasive Bladder Cancer Patients to Intravesical Bacillus Calmette-Guerin? The Role of Immunological Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Principal Investigator, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AE20121
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Bacillus Calmette-Guérin response; Prediction; Urinary cytokines; T cells; Recurrence; Progression
MeSH Terms: conditions — Urinary Bladder Neoplasms; Recurrence; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High risk NMIBC (Other): Patients with primary or recurrent NMIBC for whom primary TURBT was done and intravesical BCG was administered
  Interventions: Diagnostic Test: Urine ELISA for immunological markers (IL-2 and IL-10); Diagnostic Test: Reverse transcriptase-quantitative polymerase chain reaction (RT-qPCR) analysis

INTERVENTIONS:
Diagnostic Test: Urine ELISA for immunological markers (IL-2 and IL-10) — IL-2 and IL-10 levels were measured in the supernatants. Natural human-produced IL-2 and IL-10 concen¬trations were determined in the urine of all patients and controls by solid phase ELISA Quantikine IL-2 Immunoassay and IL-10 Immunoassay, respectively
Diagnostic Test: Reverse transcriptase-quantitative polymerase chain reaction (RT-qPCR) analysis — blood samples using QIAamp® RNA Blood Mini kit (QIAGEN, USA). 1 μg of total RNA was reverse transcribed with random primers, using High Capacity cDNA Archive Kit (Applied Biosystems, Foster City, CA, USA). RT-qPCR analysis was carried out with SYBER Green PCR Master Mix (Applied Biosystems, Foster City, CA, USA). Primers for TNF-α, CTLA4, T-bet+, GATA3+, FoxP3+ and GABDH as PCR control

SUMMARY:
Intravesical BCG is the mainstay adjuvant management of high risk NMIBC. Adequacy of immune system stimulation is the determinant factor for patient response to BCG. Immunological markers for BCG-response could be helpful for urologists especially in the era of BCG shortage.

Objectives: To assess the predictive performance of different immunological markers on BCG-response in high risk NMIBC BCG-naïve patients.

DETAILED DESCRIPTION:
Background: Intravesical BCG is the mainstay adjuvant management of high risk NMIBC. Adequacy of immune system stimulation is the determinant factor for patient response to BCG. Immunological markers for BCG-response could be helpful for urologists especially in the era of BCG shortage.

Objectives: To assess the predictive performance of different immunological markers on BCG-response in high risk NMIBC BCG-naïve patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with primary or recurrent NMIBC for whom primary TURBT was done.

Exclusion Criteria:

1. Patients with previous BCG instillation,
2. benign pathology
3. Variant histology
4. Non urothelial carcinoma,
5. concommitent upper tract urothelial tumors, detrusor muscle invasion
6. low or intermediate risk NMIBC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Initial BCG complete response | 3 months
  free cystoscopy/negative cytology at 3 months.
Recurrence | 1 year
  Recurrence is defined as development of new tumor/positive cytology in patients with ICR
Progression | 1 year
  persistent/recurrent tumor during or after treatment with increasing tumor grade or upstaging to muscle invasion after initial complete response

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Elsawy, Principal Investigator — Urology and Nephrology Center
Locations (1):
- Urology and Nephrology Center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: No